CLINICAL TRIAL: NCT04666246
Title: Inspiratory Effort Assessment in Patients With COVID-19 Pneumonia Undergoing Non Invasive Respiratory Support
Brief Title: Inspiratory Effort in COVID-19
Acronym: PERSIA
Status: Recruiting | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Roberto Tonelli, MD, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio17
Record Dates: First submitted 2020-12-11; First posted 2020-12-14 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Acute Respiratory Failure; Covid19
Keywords: Acute respiratory failure; Esophageal pressure; Non invasive respiratory support; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at assessing esophageal pressure in patients with acute respiratory failure due to COVID-19 undergoing non invasive respiratory support.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19
* Acute respiratory failure undergoing non-invasive respiratory support

Exclusion Criteria:

* Need for immediate endotracheal intubation
* Chronic respiratory diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Respiratory Intensive Care Unit of the University Hospital of Modena for acute respiratory failure due to COVID-19 pneumonia and candidate to non invasive respiratory support
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Inspiratory effort quantification | 24 hours from admission
  Esophageal pressure assessment through dedicated esophageal pressure transducer

SECONDARY OUTCOMES:
Non invasive respiratory support failure | 24 hours
  Reaching of the criteria for endotracheal intubation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No